CLINICAL TRIAL: NCT02898220
Title: Trans-MAPP Study of Urologic Chronic Pelvic Pain: Control Study Protocol
Brief Title: Trans-MAPP II Study of Urologic Chronic Pelvin Pain
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 825428; U01DK082316 (NIH)
Record Dates: First submitted 2016-08-24; First posted 2016-09-13 (Estimated); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Interstitial Cystitis; Chronic Prostatitis
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biologic specimens collected during the course of the study include urine, blood, saliva, and rectal and vaginal swabs.
Oversight: Data Monitoring Committee: No

SUMMARY:
The Multidisciplinary Approach to the Study of Chronic Pelvic Pain (MAPP) Research Network has been established by the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) of the National Institutes of Health (NIH) to focus on a broader approach to the study of Interstitial Cystitis (IC)/ Bladder Pain Syndrome (BPS) in men and women, and Chronic Prostatitis (CP)/Chronic Pelvic Pain Syndrome (CPPS) in men, than previously undertaken. Patients with IC or CP are being recruited for a new study called the "Trans-MAPP Study of Urologic Chronic Pelvic Pain: Symptom Patterns Study (SPS). This research study will recruit Control Participants to better understand the symptoms of individuals with some form of IC or CP. As with many chronic pain disorders, IC and CP are poorly understood, and treatment is often not helpful. The goal of this study is to better understand how pain is felt in people with IC or CP and the investigators hope that this study will lead to improvement in the treatment of IC and CP.

DETAILED DESCRIPTION:
Urological Chronic Pelvic Pain Syndromes (UCPPS) are characterized by pelvic pain with concurrent urinary symptoms. Broadly, UCPPS comprise Interstitial Cystitis/Painful Bladder SyndromeBladder Pain Syndrome (IC/BPS) in men and women, and Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS) in men. IC is a debilitating bladder disorder characterized by urinary urgency, frequency, and pain. The presentation of symptoms can be quite variable among patients, suggesting that IC is a multi-factorial syndrome with several proposed etiologies, some of which may be interrelated.1 BPS as defined by the International Continence Society, is "the complaint of suprapubic pain related to bladder filling, accompanied by other symptoms, such as increased daytime and night-time frequency, in the absence of proven urinary infection or other obvious pathology."2 BPS is a clinical description of disease based on the patient's symptoms, and does not depend on urodynamic or cystoscopic findings. These symptoms may be related to IC, although diagnostic criteria are still lacking for this entity, and the relationship between BPS and IC is not clear. After the initiation phase for the MAPP SPS Study, it became clear that many of the hypotheses being proposed required well-characterized healthy "normal" controls that lack urologic pain as well as other study related symptoms/conditions. This second phase is enriched with pre-defined subgroups and a longer follow-up period which will allow further investigation of clinical and biologic factors associated with worsening and/or improvement of reported urinary and non-urinary symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Participant has signed and dated the appropriate Informed Consent document.
* Agreed to participate in ALL required study procedures (including Biospecimen collections, Neuroimaging, and Quantitative Sensory Testing).
* Gave permission for use of DNA for genetics studies.
* Gender recorded in Participant Registration module.
* Participant is at least 18 years of age.
* Participant is able to speak, read, and understand English.
* Participant reports a response of "0" (zero) on the pain, pressure or discomfort scale (SYM-Q, Question #1).
* Participant reports no chronic pain in the pelvic or bladder region, and reports no chronic pain in any other body region.
* Participant reports no urological symptoms that have been evaluated, but are still present.

Exclusion Criteria:

* Participant has an on-going symptomatic urethral stricture.
* Participant has an on-going neurological disease or disorder affecting the bladder or bowel fistula.
* Participant has a history of cystitis caused by tuberculosis, radiation therapy or Cytoxan/cyclophosphamide therapy.
* Participant has augmentation cystoplasty or cystectomy.
* Participant has an active autoimmune or infectious disorder (such as Crohn's Disease or Ulcerative Colitis, Lupus, Rheumatoid Arthritis, Multiple Sclerosis, or HIV).
* Participant has a history of cancer (with the exception of skin cancer).
* Participant has current major psychiatric disorder or other psychiatric or medical issues that would interfere with study participation (e.g. dementia, psychosis, upcoming major surgery, etc.).
* Participant has severe cardiac, pulmonary, renal, or hepatic disease that in the judgment of the study physician would preclude participation in this study.
* Participant has had definitive treatment for acute epididymitis, urethritis, vaginitis.
* Participant has history of unevaluated hematuria, this will require the evaluation of a study physician to determine if this has been appropriately evaluated.
* Participant has had a cystoscopy with hydrodistention or kenalog injection.

Exclusion Criteria for Males Only:

* Diagnosis of unilateral orchalgia, without pelvic symptoms.
* History of transurethral microwave thermotherapy (TUMT), transurethral needle ablation (TUNA), balloon dilation, prostate cryo-surgery, or laser procedure.
* A prostate biopsy or transurethral resection of the prostate (TURP) within the last three months.

Exclusion Criteria for Females Only:

• Participant has a positive Urine pregnancy test.

Specimen Exclusion Criteria (Males and Females):

• Participant has a positive dipsticParticipant has a positive urine culture.

Fatigue Symptom Eligibility Criteria:

* Participant, for at least 3 months in the past year, has persistent fatigue not relieved with rest.
* Participant, for at least 3 months in the past year, has extreme fatigue following exercise or mild exertion.
* Participant, for at least 3 months in the past year, has impaired memory, concentration or attention.

Exclusion Criteria - Urine test results:

A clean-catch midstream urine specimen (VB2) will be obtained from all male and female participants during the initial and 6 month study visits, so that a urine dipstick analysis can be done for all participants, and a urine pregnancy test can be conducted for females of child bearing age excluding those who are post-menopausal and those with a history of hysterectomy.

* If participant has an abnormal dipstick urinalysis indicating abnormal levels of nitrites and/or occult blood, that in the opinion of the Principal Investigator warrants exclusion, participant will be ineligible for study participation at the initial visit and withdrawn from study participation. A positive dipstick at the 6 Month visit will also result in the participant being withdrawn.
* If participant has had a positive urine culture in the past 6 weeks, or currently has a midstream urine culture (VB2) (>100,000 CFU/ml), with a single uropathogen, the participant will be ineligible for the study at the initial visit, treated and withdrawn from study participation. A positive dipstick at the 6 Month visit will also result in the participant being treated and withdrawn. (Must be documented on Urine Culture Result - UCR form). We will keep all specimens and data collected from both eligible and in-eligible participants unless participant request that his/her data be destroyed, and not utilized for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Trans-MAPP II control study will recruit healthy controls (male and female) over a two year period.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-09; Primary Completion 2020-07 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Pain Severity Score | 6 months
  The outcome measures are the same scores which will be used to compare normal The scores for pain severity in healthy individuals with scores of those with a diseased state (i.e. individuals with UCPPS)
Urinary Severity Score | 6 months
  The outcome measures are the same scores which will be used to compare normal The scores for urinary severity in healthy individuals with scores of those with a diseased state (i.e. individuals with UCPPS

CONTACTS AND LOCATIONS:
Overall Officials: Richard Landis, Ph.D., Study Director — University of Pennsylvania; Christopher Mullins, Ph.D, Study Director — NIDDK, NIH; J. Quentin Clemens, MD, MSCI, Study Director — University of Michigan
Locations (6):
- United States (6):
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Ann Arbor, Michigan
  - Washington University, St. Louis, St Louis, Missouri
  - University of Washington, Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Plans are still to be finalized